CLINICAL TRIAL: NCT03435562
Title: Assessment of Two New Electronic Cigarettes in Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM20012013
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- electronic cigarette vs own brand use (Experimental): Participants will come in for three session. During one session, participants will first complete a 10-puff product use bout with JUUL, and then a 90-minute ad lib product use bout with JUUL (the session will be approximately 3 hours). During one session, participants will first complete a 10-puff product use bout with IQOS, and then a 90-minute ad lib product use bout with IQOS (the session will be approximately 3 hours). During one session, participants will first complete a 10-puff product use bout with their own brand cigarettes, and then a 90-minute ad lib product use bout with their own brand cigarette (the session will be approximately 3 hours). The order of the sessions will be determined randomly and data about session will not be recorded or used in the analysis.
  Interventions: Other: JUUL electronic cigarette; Other: IQOS electronic cigarette; Other: Own Brand cigarette

INTERVENTIONS:
Other: JUUL electronic cigarette — Effects of JUUL electronic cigarette use.
Other: IQOS electronic cigarette — Effects of IQOS electronic cigarette use.
Other: Own Brand cigarette — Effects of own brand cigarette use.

SUMMARY:
The purpose of this study is to determine differences in nicotine delivery, user behavior, subjective effects, and physiological effects, when cigarette smokers use an two new electronic cigarette devices (JUUL and IQOS) relative to their using their own brand of cigarettes.

ELIGIBILITY:
Inclusion Criteria--participants must be:

* healthy (determined by self-report)
* between the ages of 18-55
* willing to provide informed consent
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol
* cigarette smokers

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Individuals who weigh less than 110 pounds

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Clinical Behavioral Pharmacolgy Laboratory, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electronic Cigarette vs Own Brand Use
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Electronic Cigarette vs Own Brand Use
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 8
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Nicotine
Description: Change in plasma nicotine level
Time Frame: Blood will be taken 4 times in each session: at baseline, 5 min after the start of a 10-puff product use, and then before and after an approximately 1-hour ad lib use period.
Population: One participant was missing a sample so data was only available for 17 participants for these analyses.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- JUUL Electronic Cigarette Use: During each session, participants will first complete a 10-puff product use bout with JUUL, and then a 90-minute ad lib product use bout with JUUL (each session will be approximately 3 hours).
  JUUL electronic cigarette: Effects of JUUL electronic cigarette use.
- IQOS Electronic Cigarette Use: During each session, participants will first complete a 10-puff product use bout with IQOS, and then a 90-minute ad lib product use bout with IQOS (each session will be approximately 3 hours).
  IQOS electronic cigarette: Effects of IQOS electronic cigarette use.
- Own Brand Cigarette Use: During each session, participants will first complete a 10-puff product use bout with their own brand cigarettes, and then a 90-minute ad lib product use bout with their own brand cigarette (each session will be approximately 3 hours).
  Own Brand cigarette: Effects of own brand cigarette use.
Arm/Group | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use | Own Brand Cigarette Use
Number analyzed (Participants) | 17 | 17 | 17
ng/ml
  Post puff bout | 7.62 (4.86) | 10.65 (6.20) | 18.31 (11.39)
  Post ad lib | 7.19 (8.32) | 5.97 (7.70) | 12.23 (9.26)

2. Secondary Outcome: Carbon Monoxide Levels
Description: Carbon monoxide levels (in parts per mission)
Time Frame: Carbon monoxide levels will be assessed before and after product use in each approximately 4-hr session: at baseline, 5 min after the end of a 10-puff product use, and then before and after an approximately 1-hour ad lib use period.
Measure: Mean (Standard Deviation); unit: Parts per mission
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
Parts per mission
  Pre puff bout | 5.2 (2.4) | 5.5 (2.4) | 5.3 (2.0)
  Post puff bout | 8.7 (2.5) | 5.1 (2.3) | 4.9 (1.8)
  Pre ad lib | 8.8 (2.8) | 5.3 (2.4) | 4.6 (1.8)
  Post ad lib | 16.6 (7.0) | 4.7 (1.9) | 4.3 (1.4)

3. Secondary Outcome: Tiffany-Drobes Questionnaire of Smoking Urges - Factor 1
Description: This scale is used to assess the extent to which product use reduces the intention to smoke a cigarette, and consists of 5 items that are scored 0 - 7, in which participants clicked seven discrete ratings from 'not at all' to 'extremely'. The items are summed and scores range from 0 to 30 with higher scores indicating higher craving for a cigarette.
Time Frame: Questionnaire will be administered 4 times in each each approximately 4-hr session: before any product use, 10 minutes after the start of a 10-puff use bout, and then before and after an approximately 1-hour ad lib use period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a scale
  Pre puff bout | 24.8 (8.2) | 24.7 (7.5) | 25.1 (8.2)
  Post puff bout | 13.2 (10.7) | 20.1 (9.3) | 16.0 (9.3)
  Pre ad lib | 21.2 (8.9) | 21.7 (9.3) | 20.4 (8.5)
  Post ad lib | 11.5 (10.2) | 17.8 (10.6) | 14.4 (9.7)

4. Secondary Outcome: Tiffany-Drobes Questionnaire of Smoking Urges - Factor 2
Description: This scale is used to assess the extent to which product use reduces the intention to smoke a cigarette, and consists of 4 items that are scored 0 - 7, in which participants clicked seven discrete ratings from 'not at all' to 'extremely'. The items are summed and scores range from 0 to 24 with higher scores indicating higher craving for a cigarette.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a scale
  Pre puff bout | 11.7 (8.3) | 10.3 (8.3) | 12.5 (8.4)
  Post puff bout | 6.9 (7.4) | 8.1 (7.8) | 6.6 (7.8)
  Pre ad lib | 9.7 (7.4) | 9.5 (7.5) | 9.1 (8.6)
  Post ad lib | 5.5 (7.6) | 6.5 (7.2) | 6.6 (8.9)

5. Secondary Outcome: Hughes-Hatsukami Questionnaire - Anxious
Description: This scale is used to assess the extent to which product use affects on anxiety and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: Questionnaire will be administered 4 times in each approximately 4-hr session: before any product use, 10 minutes after the start of a 10-puff use bout, and then before and after an approximately 1-hour ad lib use period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a scale
  Pre puff bout | 46.3 (32.5) | 42.8 (31.9) | 44.5 (34.9)
  Post puff bout | 24.8 (30.6) | 24.4 (31.8) | 28.4 (33.9)
  Pre ad lib | 22.1 (22.8) | 20.8 (30.1) | 17.2 (27.2)
  Post ad lib | 19.4 (27.5) | 20.4 (27) | 28.4 (32.6)

6. Secondary Outcome: Hughes-Hatsukami Questionnaire - Craving
Description: This scale is used to assess the extent to which product use affects on craving a cigarette and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 75.2 (30.7) | 70.5 (30.9) | 73.5 (33.5)
  Post puff bout | 34.9 (35) | 49.3 (36.0) | 42.9 (31.8)
  Pre ad lib | 55.2 (30.5) | 54.0 (38) | 53.8 (29.9)
  Post ad lib | 25.5 (29.2) | 53.9 (34.9) | 36.2 (32.1)

7. Secondary Outcome: Hughes-Hatsukami Questionnaire - Depression
Description: This scale is used to assess the extent to which product use affects on depression and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 21.4 (28.3) | 15.1 (20.9) | 20.5 (26.1)
  Post puff bout | 9.8 (16.8) | 8.8 (16.6) | 15.1 (22.6)
  Pre ad lib | 11.5 (21.5) | 8.1 (17.0) | 10.6 (20.1)
  Post ad lib | 8.8 (13.6) | 8.2 (16.3) | 11.5 (21.7)

8. Secondary Outcome: Hughes-Hatsukami Questionnaire - Difficulty Concentrating
Description: This scale is used to assess the extent to which product use affects having difficulty concentrating and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 28.2 (26.4) | 37.6 (30.1) | 30.0 (31.9)
  Post puff bout | 18.5 (20.4) | 17.3 (19.9) | 24.4 (29.9)
  Pre ad lib | 18.1 (20.8) | 15.5 (22.5) | 16.8 (20.6)
  Post ad lib | 10.4 (18.1) | 17.8 (25.8) | 18.9 (27.0)

9. Secondary Outcome: Hughes-Hatsukami Questionnaire - Drowsy
Description: This scale is used to assess the extent to which product use affects feeling drowsy and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 35.2 (25) | 33.8 (28.2) | 31.9 (33.9)
  Post puff bout | 28.7 (26.1) | 21.4 (24.6) | 29.4 (26.5)
  Pre ad lib | 24.9 (24.3) | 25.9 (31.1) | 23.4 (24.6)
  Post ad lib | 23.4 (26.9) | 25.3 (27.0) | 27.4 (29.8)

10. Secondary Outcome: Hughes-Hatsukami Questionnaire - Hunger
Description: This scale is used to assess the extent to which product use affects reducing hunger and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 39.9 (22.7) | 43.2 (29.8) | 43.0 (35.5)
  Post puff bout | 31.9 (24.4) | 35.6 (33.3) | 30.2 (25.5)
  Pre ad lib | 34.8 (25.9) | 39.5 (35.9) | 37.7 (29.0)
  Post ad lib | 39.8 (30.7) | 58.4 (29.0) | 53.2 (31.9)

11. Secondary Outcome: Hughes-Hatsukami Questionnaire - Impatient
Description: This scale is used to assess the extent to which product use affects feeling impatient and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 42.1 (28.3) | 41.0 (30.6) | 51.4 (31.0)
  Post puff bout | 23.9 (27.3) | 25.9 (31.0) | 25.1 (30.9)
  Pre ad lib | 26.9 (29.3) | 31.4 (28.9) | 29.7 (30.3)
  Post ad lib | 25.5 (28.2) | 31.8 (30.5) | 27.2 (27.0)

12. Secondary Outcome: Hughes-Hatsukami Questionnaire - Irritable
Description: This scale is used to assess the extent to which product use affects feeling irritable and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 37.4 (31.0) | 34.5 (31.1) | 38.7 (33.3)
  Post puff bout | 14.9 (17.2) | 18.4 (22.1) | 19.8 (26.3)
  Pre ad lib | 14.1 (16.0) | 15.4 (22.3) | 16.8 (21.0)
  Post ad lib | 14.6 (22.0) | 15.1 (26.4) | 16.8 (24.1)

13. Secondary Outcome: Hughes-Hatsukami Questionnaire - Restless
Description: This scale is used to assess the extent to which product use affects feeling restless and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 40.8 (29.4) | 30.2 (25.5) | 28.9 (31.8)
  Post puff bout | 19.7 (24.8) | 26.9 (25.9) | 19.7 (24.6)
  Pre ad lib | 27.7 (27.2) | 17.9 (25.7) | 33.4 (31.4)
  Post ad lib | 21.5 (28.1) | 24.7 (27.6) | 27.1 (28.4)

14. Secondary Outcome: Hughes-Hatsukami Questionnaire - Desire for Sweets
Description: This scale is used to assess the extent to which product use affects having desire for sweets and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 24.2 (30.7) | 27.4 (33.3) | 24.8 (28.3)
  Post puff bout | 16.8 (21.4) | 20.3 (27.2) | 16.4 (25.7)
  Pre ad lib | 18.8 (25.8) | 20.7 (28.1) | 23.8 (27.9)
  Post ad lib | 17.9 (21.3) | 17.4 (24.0) | 20.5 (27.0)

15. Secondary Outcome: Hughes-Hatsukami Questionnaire - Urge to Smoke
Description: This scale is used to assess the extent to which product use affects having the urge to smoke and consists of 1 item scored 0 - 100 with 0 being not at all and 100 being extremely.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
points on a scale
  Pre puff bout | 76.5 (25.2) | 67.2 (29.9) | 74.7 (31.5)
  Post puff bout | 39.2 (34.8) | 48.8 (31.9) | 46.2 (29.5)
  Pre ad lib | 54.4 (27.6) | 46.9 (33.3) | 56.9 (27.8)
  Post ad lib | 24.9 (25.7) | 50.0 (31.1) | 38 (31.8)

16. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Awake
Description: One question is used to assess how much product use makes participants feel awake, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 40.9 (31.7) | 33.8 (29.9) | 36.5 (30.6)
  Post ad lib | 45.1 (31.3) | 28.1 (29.6) | 34.5 (27.4)

17. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Calm
Description: One question is used to assess how much product use makes participants feel calm, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 60.9 (36) | 47.9 (31.9) | 54.4 (31.5)
  Post ad lib | 60.7 (35.3) | 46.6 (29.7) | 43.2 (34.5)

18. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Concentrate
Description: One question is used to assess how much product use helps participants concentrate, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 34.8 (30.8) | 24.5 (26.3) | 38.5 (33.7)
  Post ad lib | 42.0 (34.3) | 27.5 (26.3) | 27.8 (27.1)

19. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Dizzy
Description: One question is used to assess how much product use makes participants feel dizzy, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 40.7 (33.4) | 33.7 (33.5) | 36.4 (33.7)
  Post ad lib | 30.1 (36.2) | 19.4 (27.2) | 26.9 (25.8)

20. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Reduce Hunger
Description: One question is used to assess how much product use reduces feeling of hunger, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 41.9 (29.9) | 35.2 (27.4) | 29.2 (28.8)
  Post ad lib | 33.0 (27.7) | 37.1 (31.0) | 34.3 (26.1)

21. Secondary Outcome: Direct Effects of Nicotine Questionnaire - Sick
Description: One question is used to assess how much product use makes participants feel sick, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 4.1 (7.5) | 8.1 (14.2) | 9.5 (19.0)
  Post ad lib | 2.6 (5.2) | 7.8 (14.4) | 10.5 (16.8)

22. Secondary Outcome: Direct Effects of Product Use Questionnaire - Pleasant
Description: A single question is used to assess if product use felt pleasant, and is scored 0 (not at all) to 100 (extremely).
Time Frame: Questionnaire will be administered 2 times in each each approximately 4-hr session: 10 minutes after the start of a 10-puff use bout, and then after an approxiamtely 1-hour ad lib use period.
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 81.4 (29.8) | 50.4 (31.6) | 58.8 (36.0)
  Post ad lib | 81.9 (24.9) | 50.6 (31.2) | 58.9 (34.4)

23. Secondary Outcome: Direct Effects of Product Use Questionnaire - Taste Good
Description: A single question is used to assess if product use tasted good, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 77.7 (29.5) | 50.5 (32.6) | 54.6 (36.4)
  Post ad lib | 74.0 (32.1) | 51.2 (30.7) | 49.8 (35.7)

24. Secondary Outcome: Direct Effects of Product Use Questionnaire - Satisfying
Description: A single question is used to assess if product use felt satisfying, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 84.3 (24.4) | 47.0 (33.2) | 58.8 (30.9)
  Post ad lib | 83.7 (24.5) | 46.5 (31.5) | 58.8 (33.3)

25. Secondary Outcome: Direct Effects of Product Use Questionnaire - Smoke Right Now
Description: A single question is used to assess if product use made them want to use the product again right now, and is scored 0 (not at all) to 100 (extremely).
Time Frame: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a question
Arm/Group | Own Brand Cigarette Use | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use
Number analyzed (Participants) | 18 | 18 | 18
score on a question
  Post puff bout | 62.8 (37.7) | 45.4 (32.7) | 47.2 (39.1)
  Post ad lib | 44.1 (37.7) | 35.5 (29.1) | 37.5 (33.5)

26. Other Pre Specified Outcome: Heart Rate
Description: Change in heart rate, measured in beats per minute
Time Frame: Heat rate will be measured from baseline continuously throughout each each approximately 4-hr session
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Blood Pressure
Description: Change in blood pressure, measured in mm/hg
Time Frame: Blood pressure will be measured from baseline continuously throughout each approximately 4-hr session
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: This protocol was minimal risk and All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | JUUL Electronic Cigarette Use | IQOS Electronic Cigarette Use | Own Brand Cigarette Use
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03435562/ICF_000.pdf
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03435562/Prot_001.pdf